CLINICAL TRIAL: NCT07314944
Title: Integrated Assessment of Sleep, Mental Health, Lifestyle Behaviors, Metabolic Markers, and Perinatal Outcomes in Women With Gestational Diabetes Mellitus: A Prospective Cohort Study
Brief Title: Maternal Sleep and Lifestyle, Metabolic Health, and Perinatal Outcomes in Gestational Diabetes
Status: Recruiting | Type: Observational
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ivana Pavlinac Dodig, Assoc Prof, University of Split, School of Medicine
Other Study IDs: 520-03/25-01/206
Record Dates: First submitted 2025-12-12; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes Mellitus; Sleep Quality; Anxiety; Mental Health; Eating Behavior; Lifestyle Factors; Physical Activity; Metabolic Markers; Glycemic Control; Perinatal Outcomes
MeSH Terms: conditions — Diabetes, Gestational; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Psychological Well-Being; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Home-Based Digital Monitoring: Pregnant women with GDM who are managed as outpatients using a short (24-36 hour) period of home-based glucose monitoring with the FreeStyle Libre system. This pathway reflects routine clinical practice for women who can return for follow-up the next day and are able to use the digital device.
  Interventions: Other: Home-Based Glucose Monitoring
- Group 2: Hospital-Based Glucose Monitoring: Pregnant women with GDM who undergo short (24-hour) inpatient glucose monitoring according to standard hospital protocols. Allocation to this pathway follows clinical logistics (e.g., distance ≥80 km, island residence) and is not assigned by the research team.
  Interventions: Other: Inpatient Glucose Monitoring

INTERVENTIONS:
Other: Home-Based Glucose Monitoring — Intervention Description: Home-Based Glucose Monitoring
  Participants undergo short-term outpatient glucose monitoring as part of routine GDM care. They follow a written schedule for capillary glucose checks while continuing normal daily activities. Data are reviewed at the follow-up visit, where routine laboratory tests and a fetal ultrasound are also performed. This approach reflects standard outpatient management for women able to return for next-day review.
  Groups: Group 1: Home-Based Digital Monitoring
Other: Inpatient Glucose Monitoring — Participants undergo a 24-hour hospital admission for scheduled capillary glucose measurements using standard hospital glucometers. During admission, participants follow the hospital's predetermined meal plan and receive continuous nursing oversight. A fetal ultrasound and routine laboratory testing are performed during the stay. This pathway follows usual clinical practice for women who require or are assigned inpatient monitoring based on logistical or clinical considerations.
  Groups: Group 2: Hospital-Based Glucose Monitoring

SUMMARY:
The goal of this observational study is to learn how sleep quality, mental health, lifestyle behaviors, and metabolic markers are related to glucose control and pregnancy outcomes in women with gestational diabetes mellitus (GDM). The main questions it aims to answer are:

* Do differences in sleep quality, anxiety levels, and eating behaviors relate to differences in glycemic control in women with GDM?
* Are maternal metabolic markers (such as glucose, liver enzymes, and lipid levels) associated with perinatal outcomes such as birth weight, cesarean delivery, and neonatal complications?
* To compare women who undergo short inpatient glucose monitoring with women who undergo home-based digital glucose monitoring to see if the mode of monitoring is related to differences in sleep, mental health, metabolic profiles, or perinatal outcomes.

Participants will:

* Complete questionnaires on sleep, anxiety, lifestyle, and eating behaviors
* Undergo routine laboratory testing, including metabolic and blood markers.
* Have glucose monitored either during a short hospital stay or through home use of the FreeStyle Libre sensor.
* Be followed from GDM diagnosis (24-34 weeks) until delivery to assess maternal and newborn outcomes

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is associated with disturbances in glucose regulation as well as a range of behavioral, psychological, and metabolic factors that may contribute to pregnancy outcomes. This prospective observational cohort study follows pregnant women with newly diagnosed GDM to evaluate how sleep quality, anxiety, eating behaviors, physical activity, and metabolic markers relate to glycemic control and perinatal outcomes.

Participants are managed according to standard clinical pathways at a tertiary obstetric center and are allocated either to short inpatient glucose monitoring or to home-based digital monitoring using the FreeStyle Libre system. These pathways reflect real-world clinical indications and are not assigned by the research team. The study leverages this natural variation to compare differences in behavioral, metabolic, and perinatal profiles between groups.

At enrollment, participants complete validated questionnaires assessing sleep quality (PSQI), anxiety (STAI), and eating behaviors (TFEQ). Clinical assessments and laboratory testing include glucose measures, liver enzymes, blood counts, and other metabolic parameters routinely collected in GDM care. Glucose monitoring data are obtained either from inpatient capillary measurements or from downloaded home-based sensor data, depending on the participant's care pathway.

Participants are followed from diagnosis (24-34 weeks of gestation) until delivery. Perinatal outcomes-including birth weight, mode of delivery, neonatal hypoglycemia, and NICU admission-are collected from medical records after delivery. The study analyzes associations between behavioral factors, metabolic markers, and both glycemic and perinatal outcomes. It also evaluates whether differences in the mode of glucose monitoring correspond to differences in maternal psychological well-being or pregnancy outcomes.

This study aims to generate multidimensional insights that may inform more personalized and less burdensome care models for women with GDM, integrating behavioral, metabolic, and clinical information to improve maternal and neonatal health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older
* New diagnosis of gestational diabetes mellitus (GDM) according to IADPSG criteria
* Gestational age 24-34 weeks at enrollment
* Able to complete study questionnaires (sleep, anxiety, eating behavior, lifestyle)
* Able to provide informed consent
* For participants in the home-monitoring pathway: ability to use a smartphone and the FreeStyle Libre device

Exclusion Criteria:

* Pre-existing type 1 or type 2 diabetes mellitus
* Current preeclampsia or major obstetric complications at enrollment
* Major psychiatric disorders interfering with participation
* Chronic use of sedatives or anxiolytic medications
* Inability to complete questionnaires
* Planned delivery outside the study's hospital network
* Any condition judged by clinicians to interfere with participation or data reliability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged 18 years or older with a new diagnosis of gestational diabetes mellitus (GDM) between 24 and 34 weeks of gestation who are receiving routine antenatal care at a tertiary obstetric center. Participants represent a real-world clinical population managed either with short inpatient glucose monitoring or home-based digital monitoring, depending on standard clinical pathways. The study population includes women able to complete questionnaires on sleep, mental health, and lifestyle behaviors and willing to participate until delivery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Perinatal Outcome | At delivery/birth
  Proportion of participants experiencing any of the following outcomes in the newborn: macrosomia (birth weight ≥4000 g), neonatal hypoglycemia requiring intervention, admission to neonatal intensive care unit (NICU), 5-minute Apgar score <7, or stillbirth.

SECONDARY OUTCOMES:
Sleep Quality (PSQI Score) | At enrollment (24-34 weeks of gestation)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated self-administered questionnaire consisting of 19 items that generate a global score ranging from 0 to 21, as well as seven component (subscale) scores.
  The global PSQI score (range 0-21) and individual component scores will be analyzed as continuous variables. Higher PSQI scores indicate poorer sleep quality, while lower scores reflect better sleep quality.
Anxiety Levels (STAI Score) | At enrollment (24-34 weeks of gestation)
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI), a validated self-report instrument comprising two 20-item subscales: STAI-State (situational anxiety) and STAI-Trait (general anxiety proneness).
  Each subscale yields a score ranging from 20 to 80, analyzed as a continuous measure. Higher STAI scores indicate greater anxiety, whereas lower scores indicate lower anxiety levels.
Eating Behaviors (TFEQ Subscales) | At enrollment (24-34 weeks of gestation)
  Eating behaviors will be assessed using the Three-Factor Eating Questionnaire (TFEQ), a validated self-report instrument that evaluates three domains of eating behavior: cognitive restraint, uncontrolled eating, and emotional eating.
  Each TFEQ subscale is scored according to the instrument's standard scoring procedure and analyzed as a continuous measure. Higher scores on each subscale indicate a greater degree of the corresponding eating behavior (i.e., greater cognitive restraint, greater uncontrolled eating, or greater emotional eating), whereas lower scores indicate a lesser degree of that behavior.
Mean Glucose Level | During the 24-36 hour monitoring period (home or inpatient)
  Average interstitial or capillary glucose level obtained from sensor downloads or hospital measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive pregnancy-related clinical, psychological, and metabolic data, and current approvals cover analysis only within the research team. De-identified, aggregate data may be shared in publications or upon reasonable request.